CLINICAL TRIAL: NCT02539979
Title: A Double Blinded Randomized Control Trial of Intravenous Paracetamol vs. Placebo in Patients Receiving Radiofrequency Ablation of the Medial Branch Facet Nerve
Brief Title: A Trial of Intravenous Paracetamol vs. Placebo in Patients Receiving Radiofrequency Ablation of the Medial Branch Facet Nerve
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Matthew Medwick, MD, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2351-15
Record Dates: First submitted 2015-09-01; First posted 2015-09-03 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Chronic Lower Back Pain; Lumbar Facet Syndrome
Keywords: IV Paracetamol; Radiofrequency Lesion/Ablation of medial branch nerve; Preventative Pain Management
MeSH Terms: interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- IV Paracetamol (Active Comparator): Patients will receive 1gram of IV paracetamol mixed in 100ml infused over 15 minutes. The patients will undergo radiofrequency lesioning of two consecutive levels of lumbar facets under fluoroscopic guidance
  Interventions: Drug: Paracetamol
- IV Placebo (Normal Saline) (Placebo Comparator): Patients will receive 100ml of normal saline infused over 15 minutes. The patients will undergo radiofrequency lesioning of two consecutive levels of lumbar facets under fluoroscopic guidance
  Interventions: Drug: Placebo - Normal Saline

INTERVENTIONS:
Drug: Paracetamol
  Arms: IV Paracetamol
Drug: Placebo - Normal Saline — Normal Saline 100cc
  Arms: IV Placebo (Normal Saline)

SUMMARY:
A double blinded randomized controlled study comparing pre-procedural IV Paracetamol versus IV placebo (normal saline). The patients will be randomized to either receiving IV paracetamol or saline infusions before undergoing radiofrequency lesioning of two levels of medial branch nerves of the lumbar facets. The primary outcome will be potential differences in pain control. The secondary outcomes will be changes in quality of life (QoL) and activities of daily living (ADLs). We will also be comparing potential differences in the amounts of post-procedure pain medications taken by the patients in each wing of the study

DETAILED DESCRIPTION:
The experiment will take place in the Chaim Sheba TelHashomer Medical Center, Tel Aviv, Israel. Patients will be recruited from the hospital's Pain Management outpatient facility from those appropriate for the procedure involving Radiofrequency Ablation of the Medial Branch of the Facet Nerve. After receiving the hospital's Helsinki approval, the P.I. and/or other designated staff in the department will approach relevant patients (in line with the mentioned inclusion and exclusion criteria), describe the procedure, and collect informed consent if the patient is interested in participating. Consent will be obtained from the patient during the patient visit when the option of RF is agreed upon and scheduled for the future.

Subjects will not receive any monetary compensation. It will be stressed to prospective subjects that participation in the research will not have any implications on their treatment in the hospital, or the relationship with their current healthcare providers. The patients will be advised that they may unconditionally revoke their consent at any given time during participation without repercussion on future care. Pt will be advised that they may withdraw from participation at any time. Data collected during the experiment will be kept in a secure location and will be shredded after the project's completion. All information regarding patient treatment both inside and outside of the project will be kept in the utmost of confidentiality, respecting both legal and ethical constraints.

Patients will be double-blindedly assigned to either IV Paracetamol or Placebo group when they arrive for their normally scheduled appointment for Radiofrequency ablation of the Median Branch Facet Nerve. Both randomization and the blinding will be done by the pharmacy of Tel Hashomer. Paracetamol will also be stored and procured from the Tel Hashomer pharmacy. Patients will be advised that neither the medical staff nor they themselves will know which they are receiving. Patients will receive a slow-infusion of either Placebo ( normal saline) or IV Paracetamol 1 g/100 ml solution over a period of 15 minutes prior to the start of the procedure. During this stage the patient will be monitored, initial VAS score recorded, and pre-operative vital signs assessed (e.g.- B/P, HR, SO2.) The same parameters will be recorded during the RF as well.

All saline bags will be numbered, mixed, and hung by one of the nurses working in the preprocedure/admission area of the pain department. The nursing staff will hold the log book containing the numbered IV infusion which each patient receives, to be recorded on the patients record for future reference. The treating physician, circulating nurse, and the patient will not have any knowledge as to whether the patient is receiving Paracetamol or Placebo.

The patient will enter the procedure room to undergo radiofrequency ablation once the infusion of IV Paracetamol/Placebo is completed. The patient will sign consent for the procedure. The patient will be placed in the prone position. The area of skin over which the procedure will be performed will be prepared and draped in standard sterile fashion. 1.5cc of Midazolam will be given for lite anesthesia. Fluoroscopy will be used to identify the specific site of the injections and radiofrequency. Lidocaine 1% will be inject to the site of the procedure to provide local anesthesia. Radiofrequency probe needles will be place to the determined medial branches under fluoroscopic guidance, with confirmation of placement established by electrical parameters. The a dilution of 2cc Lidocaine 1% 1cc and Depomedrol 40mg will be injected prior to ablation of each nerve. Ablation of the nerve will be conducted with thermal heat of 80 degrees Celsius for one minute for each nerve. 3cc solution of Lidocaine 1% + Depomedrol 40mg will be injected around each nerve after the ablation has been performed. A sterile bandage will be placed over the needle entry points, and the patient will be transferred to the recovery area for further monitoring.

Following the procedure the patient will be taken to the recovery room in the pain clinic and will be monitored for 30 minutes. Vitals will be assessed immediately post-op in the recovery room and again after 30 minutes, just prior to discharge. They will be asked when they get to the recovery room and again after 30 minutes, prior to discharge, to assess their level of pain. Requests for additional analgesia (Optalgin, etc) will be assessed. Pt will be asked at 0 minutes and at 30 minutes following entry to recovery room if they are experiencing any of a number of side effects and there responses noted in their records.

Patients will be provided with a packet containing copies of the Oswestry and Roland Disability Questionaires. The patients will complete both questionaires daily (at noon) for the first week and then weekly for the remaining 5 weeks of follow up. The questionnaire evaluate the patients' pain level, level of functioning, and measures of quality of life.

All patients will be seen for follow up appointment with their treating pain physician in the Pain Department of Tel HaShomer 6 weeks following the procedure. Patients will return with their journals and will have their vitals, pain assessment score, and other symptoms (if any) assessed once more at the final visit.

Results A comprehensive review and statistical analysis of data will be conducted at the completion of the study. Changes in pain scores, as reported by the patients via the VAS scores, will be analyzed as change in pain score over time. Cumulative VAS scores for each group will be compared using the Mann-Whitney U-test and the t-test. Changes in ADL and QoL will be measure using the Roland Disability Questionnaire and the Oswestry low back pain disability scales. Both the Roland Disability Questionnaire and the Oswestry scores will be completed by the patients both before the procedure and at the six week completion. Results from both will be statistically analyzed with the Mann-Whitney U-test and by t-test.

ELIGIBILITY:
Inclusion Criteria:

* • Men and women.

  * Age of 18+ years
  * Weight over 50 kg
  * Fits criteria for procedure-- radiofrequency ablation of medial branch facet nerve

Exclusion Criteria:

* • Patients who are incapable of judgment and\or to give informed consent.

  * Pregnant or nursing.
  * Under 18 years old
  * Allergies to Paracetamol, Lidocaine, Midazolam, Depomerol
  * Chronic Paracetamol use (or products with Paracetamol- e.g.- Zaldiar) 2 weeks preoperatively.**
  * Chronic NSAID use (or products containing NSAIDS) for 2 weeks pre-operatively.**
  * Illicit Drug use 48 hours prior to participation.
  * Current alcohol abuse (3 or more alcoholic drinks per day)
  * Severe liver disease
  * Severe cardiac disease
  * Severe renal disease
  * Platelet dysfunction or other bleeding disorder
  * Currently unstable psychiatric disorders.
  * Primary diagnosis of fibromyalgia
  * **If the patient is taking chronic pain medication other than Paracetamol or NSAIDS they may continue to take them and it will be standardized and accounted for (eg.- opioids to morphine mEq).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-08; Primary Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Pain Reduction | 6 weeks
  To examine the potential impact of intravenous paracetamol on the level of pain during the 6 weeks following radiofrequency of the medial branch facet nerve

SECONDARY OUTCOMES:
Change in demand for pain medication | 6 weeks
  To examine the potential reduced need for additional analgesia in the 6 weeks following radiofrequency of the medial branch facet nerve

OTHER OUTCOMES:
Quality of Life and Activities of Daily Living | 6 weeks
  To examine potential changes in quality of life measures with pre-procedure IV paracetamol

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel, Israel